CLINICAL TRIAL: NCT07053722
Title: Observational Clinical Study of Patients With Muscle - Invasive Bladder Cancer Undergoing Bladder Preservation Therapy After Neoadjuvant Therapy
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Shangbin QIN, Doctor, Peking University First Hospital
Other Study IDs: NA-TMT-001
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Bladder (Urothelial, Transitional Cell) Cancer
Keywords: radiation oncology; bladder cancer; TMT
MeSH Terms: conditions — Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NA-TMT: Patients with Muscle - Invasive Bladder Cancer Undergoing Bladder Preservation Therapy After Neoadjuvant Therapy
  Interventions: Radiation: NA-TMT

INTERVENTIONS:
Radiation: NA-TMT — After neoadjuvant therapy, patients choose trimodality therapy (TMT) for bladder preservation over radical cystectomy.

SUMMARY:
The goal of this observational study is to evaluate the safety and efficacy of neoadjuvant therapy followed by bladder - preserving TMT in patients with MIBC. The main question it aims to answer is: Does this treatment model improve long - term outcomes, including survival, local control, distant metastasis, and bladder preservation rates? Participants who received neoadjuvant therapy and underwent TMT for bladder preservation will be observed.

ELIGIBILITY:
Inclusion Criteria:

Histopathologically confirmed bladder cancer (T2-T4aN0-2M0, 8th edition AJCC staging).

Underwent bladder - sparing TMT following neoadjuvant therapy (ADC, immunotherapy, or chemotherapy).

Aged ≥18 years. Signed an informed consent form. Good general condition with ECOG performance status of 0-2. Adequate organ function for chemoradiotherapy: (1) Hematology: Absolute neutrophil count ≥1.5×10⁹/L, platelets ≥100×10⁹/L, hemoglobin ≥90 g/L. (2) Liver function: Total bilirubin ≤1.5×ULN, ALT and AST ≤2.5×ULN (≤5×ULN if hepatic metastasis is present). (3) Renal function: Creatinine clearance ≥30 mL/min (via Cockcroft-Gault formula).

Exclusion Criteria:

Distant metastasis (M1). Other malignancies (except cured basal cell carcinoma or cervical carcinoma in situ).

Severe cardiovascular disease (uncontrolled heart failure, unstable angina, myocardial infarction, etc.).

Severe hepatic/renal dysfunction intolerance to chemoradiotherapy. Mental illness/cognitive impairment unable to comply with the study. Allergy to chemoradiotherapy drugs. Pregnant or breastfeeding women. Previous pelvic radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histopathologically confirmed bladder cancer (T2-T4aN0-2M0, 8th edition AJCC staging).
  Underwent bladder - sparing TMT following neoadjuvant therapy (ADC, immunotherapy, or chemotherapy).
  Aged ≥18 years. Signed an informed consent form. Good general condition with ECOG performance status of 0-2. Adequate organ function for chemoradiotherapy: (1) Hematology: Absolute neutrophil count ≥1.5×10⁹/L, platelets ≥100×10⁹/L, hemoglobin ≥90 g/L. (2) Liver function: Total bilirubin ≤1.5×ULN, ALT and AST ≤2.5×ULN (≤5×ULN if hepatic metastasis is present). (3) Renal function: Creatinine clearance ≥30 mL/min (via Cockcroft-Gault formula).
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
DFS | 5 years
OS | 5 years
BI - EFS | 5 years

IPD SHARING:
Plan to Share IPD: Undecided